CLINICAL TRIAL: NCT03568799
Title: [18F] 4-L-Fluoroglutamine (2S,4R) PET/CT in Imaging Patients With Newly Diagnosed Lung Cancer or Indeterminate Pulmonary Nodules
Brief Title: 4-[18F]Fluoroglutamine PET/CT in Imaging Patients With Newly Diagnosed Lung Cancer or Indeterminate Pulmonary Nodules
Acronym: GLN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XH-17-012
Record Dates: First submitted 2017-12-13; First posted 2018-06-26 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer; Solitary Pulmonary Nodule; Cigarette Smoking Behavior
MeSH Terms: conditions — Lung Neoplasms; Solitary Pulmonary Nodule; Cigarette Smoking | interventions — 4-fluoroglutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-[18F]Fluoroglutamine (Experimental): Patients undergo 18F-FDG PET/CT scan first. Within 7 working days, patients receive 4-[18F]Fluoroglutamine IV and 60 minutes after injection, undergo 4-[18F]Fluoroglutamine PET/CT before the start of therapy.
  Interventions: Radiation: 18F-(2S,4R)4-fluoroglutamine

INTERVENTIONS:
Radiation: 18F-(2S,4R)4-fluoroglutamine — Undergo 18F-(2S,4R)4-fluoroglutamine PET/CT

SUMMARY:
This clinical trial studies positron emission tomography (PET) imaging utilizing 18F-(2S,4R)4-fluoroglutamine, a glutamic acid derivative, to image patients with Newly Diagnosed Lung Cancer or Indeterminate Pulmonary Nodules. [18F]Fluoroglutamine PET may provide additional information that help diagnose lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients are given the opportunity to participate in the study if

  1. Age between 18-79;
  2. The patient must be able to give informed consent;
  3. Sexually active subjects agree to use condoms and/or their partners of reproductive potential to use a method of effective birth control during imaging period of 2 weeks;
  4. Patients can finish PET/CT scan without tranquilizers;
  5. Patients with a newly diagnosed, untreated primary lung cancer; Or patients older than 55, current or former smoking with ≥ 30 pack years, and newly discovered indeterminate pulmonary nodules (7-30 mm diameter) on CT.
  6. No chemotherapy, radiotherapy or immune/biologic therapy,or biopsy were allowed between the 18F-FDG and the 4-[18F]Fluoroglutamine PET/CT.

Exclusion Criteria:

* Patients with any of the following conditions will be excluded

  1. Pregnant or lactating patients;
  2. Patients with active lung infection;
  3. Inability or refusal to have at least one peripheral intravenous line for intravenous access;
  4. From assays obtained <2 weeks prior to study enrollment（ULN：the upper limit of normal value ）:Bilirubin>1.5*ULN,AST/ALT >2.5 * ULN, Albumin< 3 g/dl, GGT > 2.5 x ULN if ALP> 2.5 x ULN, Creatinine>1.5*ULN or creatinine clearance <60ml/min；
  5. Patients with a history of allergic reaction to this drugs or its analogues；
  6. patients with poor compliance;
  7. Acute major illness

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosing and Staging ability of 4-[18F]Fluoroglutamine PET/CT in lung cancer | up to three years
  Sensitivity, specificity, diagnostic accuracy of 4-[18F]Fluoroglutamine and 18F-FDG PET/CT will be compared using paired t-test or Krusal-Wallis test.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 30 days after the F-Gln imaging
  The evaluation of the Incidence of Treatment-Emergent Adverse Events starts from the day of F-Gln examination until 30 days later; Treatment-Emergent Adverse Events are evaluated according to version 4.03 CTC-AE criteria.
ASCT2 expression levels in tissue samples | up to three years
  Wilcoxon rank-sum or Kruskal-Wallis tests will be applied for the group comparisons of IHC staining(ASCT2)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided